CLINICAL TRIAL: NCT00496951
Title: Vagal Tone and Neonatal Abstinence Syndrome
Acronym: NAS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 6468; R01DA019934 (NIH)
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Neonatal Abstinence Syndrome; Vagal Tone
Keywords: Neonatal abstinence syndrome; Methadone; Vagal tone
MeSH Terms: conditions — Neonatal Abstinence Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vagal tone assessment — An EKG will be obtained using a Physio-control EKG monitor (R wave Electronics of Florida) in standard application, with three chest leads. The EKG data is inputted into a vagal tone monitor (Delta Biometrix, Bethesda MD) which computes vagal tone from the EKG signal. This data is then transferred to a disk which is analyzed off-line.
  Other Names: EKG monitor (R wave electronics); Vagal tone monitor (Delta Biometrix)

SUMMARY:
Symptoms of Neonatal Abstinence Syndrome (NAS) can be attributed largely to dysfunction of the autonomic nervous system in opiate exposed neonates. Vagal tone is a readily available measure of autonomic nervous system functioning. NAS is a widely variable disorder with poorly understood pathophysiology; while all opiate exposed infants will exhibit some signs and symptoms of NAS, only approximately ½ have severe enough symptoms to require pharmacologic therapy. This research seeks to determine the relationship between infant vagal tone and NAS severity. The determination of a link between newborn vagal tone and NAS severity could result in the prediction of infants at risk for severe NAS and provide these infants and mothers with intensified services and early treatment, thereby shortening the course of NAS in the infant.

DETAILED DESCRIPTION:
Consecutively born methadone exposed infants had hert period and cardiac vagal tone measurements extracted via standard EKGs on days 1 and 3 of life. The infant's NAS course was assessed serially.

ELIGIBILITY:
Inclusion Criteria:

* Term infant (>= 37 weeks by 1st or second trimester sonogram),
* In utero opiate exposure (either heroin or methadone) requiring a minimum of three day infant hospitalization after birth
* Delivery to a client active in drug abuse treatment

Exclusion Criteria:

* Significant medical complications in the infant
* Circumcision within 24 hours of the proposed EKG/vagal tone measurement (circumcision has been found to affect vagal tone)
* Infant hospitalization in the Neonatal Intensive Care Unit (NICU)
* Psychiatric impairment of the mother such that informed consent is not possible

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Drug exposed infants
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Jansson, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Jansson LM, Dipietro JA, Elko A, Velez M. Infant autonomic functioning and neonatal abstinence syndrome. Drug Alcohol Depend. 2010 Jun 1;109(1-3):198-204. doi: 10.1016/j.drugalcdep.2010.01.004. Epub 2010 Mar 1. PMID 20189732